CLINICAL TRIAL: NCT05667740
Title: A Phase 1, Randomised, Placebo-controlled, Double-blind, Sequential Ascending-dose Study to Evaluate the Safety, Tolerability, and Immunogenicity of an Inactivated Whole-cell Pneumococcal Vaccine (Gamma-PN3) in Healthy Adults
Brief Title: Safety, Tolerability and Immunogenicity of an Inactivated Whole-cell Pneumococcal Vaccine Gamma-PN3.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GPN Vaccines (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GPNV-001
Record Dates: First submitted 2022-12-19; First posted 2022-12-29 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2023-02

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — 13-valent pneumococcal vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Gamma-PN3 (Experimental): Inactivated whole-cell pneumococcal vaccine at 50, 250 or 1000 mcg of protein content.
  One dose on Day 1 and second dose Day 29
  Interventions: Biological: Gamma-PN3
- Placebo (Placebo Comparator): Saline on Day 1 and second dose Day 29
  Interventions: Drug: Placebo
- Prevenar-13 (Active Comparator): Licensed pneumococcal vaccine on Day 1 and saline on Day 29
  Interventions: Biological: Prevenar-13
- Pneumovax-23 (Active Comparator): Licensed pneumococcal vaccine on Day 1 and saline on Day 29
  Interventions: Biological: Pneumovax-23

INTERVENTIONS:
Biological: Gamma-PN3 — Inactivated whole-cell pneumococcal vaccine
  Arms: Gamma-PN3
Biological: Prevenar-13 — Licensed polysaccharide conjugate pneumococcal vaccine
  Arms: Prevenar-13
Biological: Pneumovax-23 — Licensed polysaccharide pneumococcal vaccine
  Arms: Pneumovax-23
Drug: Placebo — Saline
  Arms: Placebo

SUMMARY:
This is a randomised placebo-controlled first-in-man dose-ranging study to determine safety and markers of efficacy.

DETAILED DESCRIPTION:
The study is of double-blind; parallel groups dose escalation design. In each cohort of 39 participants 30 will receive Gamma-PN3; 3 will receive Prevenar; 3 will receive Pneumovax and 3 saline placebo.

The doses of Gamma-PN3 will be 50mcg; 250 mcg and 1000 mcg of protein content.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female volunteers aged 50 to 69 years inclusive at Screening.
2. In good health as determined by the outcome of medical history, physical examination, and clinical judgement by the Investigator. Chronic stable non-inflammatory conditions such as hypertension, hyperlipidemia, well-controlled type 2 diabetes, stable asthma, controlled psychiatric conditions such as anxiety or depression, stable ischemic heart disease without heart failure are permitted, as determined by the Investigator.
3. Willing and able to give voluntary written informed consent before screening assessments commence.
4. Vital signs within the following ranges (inclusive):

   * Body temperature 35.5 to 37.7°C
   * Heart rate 50 to 100 beats per minute
   * Respiratory rate 12 to 22 breaths per minute
   * Systolic blood pressure 90 to 160 mmHg
   * Diastolic blood pressure 50 to 95 mmHg
5. 12-lead electrocardiogram (ECG) parameters within the following ranges:

   * QTcB & QTcF - males ≤450 msec. females ≤470 msec
   * PR 100 to 240 msec inclusive
   * HR 50 to 100 bpm inclusive
6. Willing and able to communicate with the Investigator and study team and understands the requirements of the study.
7. Willing and able to undertake the study visits and all assessments, including possessing a suitable device and access to the internet for using the web-based electronic diary (e.g., smartphone, tablet, or computer) and able to use the device for this purpose.
8. Vaccinated against severe acute respiratory syndrome corona virus 2 (SARS-CoV-2; COVID-19) as per State Health advice at the time of recruitment.

Exclusion Criteria:

1. History of a previous Pneumovax 23® vaccination.
2. History of a previous Prevenar 13® vaccination.
3. Splenectomy or cochlear implant, due to likelihood of having received pneumococcal vaccination at age less than 70 years.
4. Positive serology blood test for human immunodeficiency virus (HIV) antibodies, hepatitis B virus (HBV) surface antigen or Hepatitis C virus (HCV) antibodies.
5. Infectious disease including but not limited to COVID-19 and influenza within 30 days before Screening and any time between Screening and Day 1 first dose, as this may confound immune response to study vaccine.
6. Liver function tests (including aspartate aminotransferase [AST], alanine aminotransferase [ALT], bilirubin) >1.5 upper limit of normal (ULN).
7. Clinically significant abnormalities in laboratory tests (biochemistry, haematology, coagulation, urinalysis), physical examination, 12-lead ECG or vital signs during the Screening period that, in the opinion of the Investigator, would affect immune response to vaccination and/or ability to fully participate in the study and/or not be in the individual's best interest to participate in the study. One retest per abnormality is permitted.
8. Participation in another clinical study of any investigational or licensed product (including investigational COVID-19 vaccines, drugs, medical devices) or medical procedure within 4 weeks from last study visit before screening.
9. Plan to have a vaccine during the study period including COVID-19 booster.
10. Have had a live vaccine within three months of the first dose of study product or any other vaccine (including any COVID-19 vaccine) within 28 days of the first dose of study product. Examples of live vaccines include, but are not limited to the following: measles, mumps, rubella, chicken pox/zoster, monkeypox, yellow fever, rabies, Bacillus Calmette-Guérin, and typhoid (oral) vaccines. Seasonal influenza vaccines for injection are generally killed virus vaccines and are permitted if administered at least 28 days before the first dose of study treatment and not during the enrollment or the study period. However, intranasal influenza vaccines are live attenuated vaccines and are not permitted within three months of first dose.
11. Have received blood or blood-derived products in the last three months before screening, which might interfere with assessment of the immune response.
12. Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the last six months before screening; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than two consecutive weeks within the last month before screening, depot or intraarticular steroids within 3 months before screening).
13. A systemic inflammatory condition such as rheumatoid arthritis or inflammatory bowel disease.
14. History of severe allergic reaction e.g., severe cutaneous adverse reaction or anaphylaxis to any medicinal product or to any of the study products, including excipients.
15. Current alcohol abuse (> 21 U/week for men and 14 U/week for women), substance dependence including nicotine/tobacco smoking (defined as more than 5 cigarettes or tobacco/nicotine equivalent per day; smoking or vaping will not be permitted while at the study unit), any use of illicit drugs or other addiction which might interfere with the ability to comply with study procedures in the opinion of the Investigator, positive drugs of abuse screen (tricyclic antidepressants are not exclusionary if consistent with medical history) or positive alcohol breath test at Screening or pre-dose. One re-test permitted for drugs of abuse screen where justified (e.g., false positive suspected).
16. Clinically significant chronic illness that, in the opinion of the Investigator, is at a stage where it might interfere with study conduct or completion. Examples include congestive heart failure, COAD with breathlessness interfering with daily activities; psychiatric conditions, poorly controlled asthma, or diabetes
17. Any chronic medical condition e.g., asthma, gout, which is likely to need systemic corticosteroid therapy during the study. -

Ages: 50 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2023-10-08 (Actual); Study Completion 2023-10-08 (Actual)

PRIMARY OUTCOMES:
Adverse events and clinical laboratory measures | 57 days
  Safety
Immunogenicity | 57 days
  Frequency of participants with > 4 fold increase in IgG titre at 29 and 57 days.

SECONDARY OUTCOMES:
OPKA response | 57 days
  Opsonophagocytic antibodies effective against different serotypes of Streptococcus pneumoniae will be assessed at Days 29 and 57

CONTACTS AND LOCATIONS:
Overall Officials: Sepehr Shakib, MD, Principal Investigator — CMAX
Locations (1):
- CMAX, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No